CLINICAL TRIAL: NCT01455558
Title: Safety and Pharmacokinetic Comparison of Cilostazol SR and IR Formulations in Healthy Korean Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Kyungsoo Park, Associate Professor, Severance Hospital
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PCF_PP-101
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Pharmacokinetics

ARMS (1):
- Cilostazol (Experimental)
  Interventions: Drug: Pletaal

INTERVENTIONS:
Drug: Pletaal — Part 1: a single dose of the SR (200mg x 1 tablet, QD) and IR (100mg x 2 tablets, BID) formulation of cilostazol orally 7 days apart in a fasted state
  Part 2: a single dose of the SR (200mg x 1 tablet, QD) formulation of cilostazol 7 days apart in a fasted and a fed state
  Part 3: multiple doses of the two formulations for eight consecutive days 21 days apart

SUMMARY:
This study investigates safety and pharmacokinetic comparison of Pacific Pharma's PP-101 SR (test formulation) and Otsuka's Pletaal® IR (reference formulation) for single and multiple doses and food effects on Pacific Pharma's PP-101 SR in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers between the ages of 19 and 55 and within 20% of their ideal body weight, without congenital abnormality or chronic disease
* Female subjects showing positive results on a serum pregnancy test before the study, and those who were of childbearing potential agreed to use one of the following medically accepted methods of contraception during the entire period of the study: abstinence, documented tubal ligation at least 1 year before enrollment in the study, documented placement of an intrauterine device with a proven failure rate of <1% per year, or double barrier methods (a spermicide plus a male condom or female diaphragm).

Exclusion Criteria:

* History of cardiovascular, pulmonary, renal, endogenous, gastrointestinal, hematologic, neurologic or hemorrhagic disease;
* Clinically significant findings on routine laboratory (hematology, serum chemistry and urinalysis) or ECG tests;
* Use of prescription drugs in the 14 days immediately prior to starting the study that had the potential to interact with the study medication;
* Use of any substance that could induce CYP3A4 synthesis (eg, St. John's wort, other herbal medications).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 0, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose for test drug; 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 18, 20, 22, 24, 36, 48, 72 hours post-dose for reference drug
  Cmax, Area Under Curve

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee D, Lim LA, Jang SB, Lee YJ, Chung JY, Choi JR, Kim K, Park JW, Yoon H, Lee J, Park MS, Park K. Pharmacokinetic comparison of sustained- and immediate-release oral formulations of cilostazol in healthy Korean subjects: a randomized, open-label, 3-part, sequential, 2-period, crossover, single-dose, food-effect, and multiple-dose study. Clin Ther. 2011 Dec;33(12):2038-53. doi: 10.1016/j.clinthera.2011.10.024. Epub 2011 Nov 29. PMID 22129569